CLINICAL TRIAL: NCT05529511
Title: The PreOperative Management of Patients Awaiting Anterior Cruciate Ligament Reconstruction: a Mixed-methods Study
Brief Title: The PreOperative Management of Patients Awaiting Anterior Cruciate Ligament Reconstruction
Acronym: POP-ACLR
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: Health Education England, Wessex (Other); University of Nottingham (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: UHDB/2020/022
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1 - Preoperative: Interviews to be completed with approximately 12 participants at three time points:
  1. Prior to anterior cruciate ligament surgery
  2. 3-month after anterior cruciate ligament surgery
  3. 12-months anterior cruciate ligament surgery
  Interventions: Other: Phase 1 - semi-structured interviews
- Phase 2 - Nominal Group Technique panel: Consensus meeting with up to 12 participants (clinicians, patients and stakeholders) to develop the prehabilitation intervention
  Interventions: Other: Phase 2 - consensus meeting

INTERVENTIONS:
Other: Phase 1 - semi-structured interviews — Semi-structured face-to-face or virtual interviews.
  Groups: Phase 1 - Preoperative
Other: Phase 2 - consensus meeting — Face-to-face or virtual meeting(s)
  Groups: Phase 2 - Nominal Group Technique panel

SUMMARY:
Patient experiences of the NHS ACL treatment pathway are unknown.

This study aims to explore patient experiences of anterior cruciate ligament ruptures at three different time points on the patient pathway: (1) 12 participants up to 2 weeks before surgery, (2) 12 participants 3 months after surgery, (3) 12 participants 12 months after surgery.

DETAILED DESCRIPTION:
The anterior cruciate ligament is one of four key ligaments in the knee. It is the most commonly injured knee ligament with an estimated 200,000 injuries occurring each year in the US (UK data unavailable). Surgery is currently standard treatment for this injury and helps patients return to work and their preinjury activity levels (such as running, playing football or netball). Patients expect surgery to be successful. However, the number of patients who are able to return to their normal activities is low, with only 24% returning at 1 year after surgery. Research has shown that after surgery, patients lack confidence, feel fearful about reinjuring their knee and need to continue to seek advice from healthcare professionals.

Receiving physiotherapy before surgery (called 'prehabilitation') is recommended by researchers and physiotherapists to help patients prepare for surgery and postoperative rehabilitation. Although physiotherapy is recommended, some patients don't receive any treatment before their operation, but it is not known why this might be. There are also no guidelines for the treatment patients receive and current treatment varies.

If an intervention to be delivered to patients prior to anterior cruciate ligament surgery (prehabilitation treatment package) is developed, patient care may be improved. Patient outcomes could also be improved resulting in more patients returning to physical activity after surgery.

This study will firstly, interview participants at three different time points along the patient pathway (1) 12 participants up to 2 weeks before surgery, (2) 12 participants 3 months after surgery, (3) 12 participants 12 months after surgery.

The interviews will allow participants to tell the story of their experiences from the point of receiving their injury diagnosis to returning to physical activity and what they expect from their surgery.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

1. ≥ 18-years-old
2. Patient who is awaiting or has previously had an ACLR in the NHS

Phase 2

1. ≥ 18-years-old
2. Participants will be in one of the following categories:

   1. Healthcare professional in the NHS with a special interest/expertise in treating ACL injuries (must have treated a patient prior to or post ACLR within the last 2 years)
   2. Therapy manager of an NHS musculoskeletal outpatient therapy department
   3. Patient who is awaiting or has previously had an ACLR in the NHS

Exclusion Criteria:

Phase 1:

1. Concomitant injuries requiring surgical intervention that will significantly alter the postoperative rehabilitation protocol e.g. meniscal repair requiring a non-weight bearing period
2. Previous knee surgery to the affected limb
3. Co-existing injuries requiring surgical intervention impacting on the individual's participation in pre-or post-operative rehabilitation
4. Pregnancy

Phase 2:

(1) Anyone with a recognised conflict of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 1: Patients who have had or who are awaiting an anterior cruciate ligament reconstruction in the NHS
  Phase 2: Healthcare professional with a special interest/expertise in treating ACL injuries, therapy manager of an NHS musculoskeletal outpatient therapy department or patient who is awaiting or has had an anterior cruciate ligament reconstruction in the NHS
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Carter, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust / University of Nottingham
Locations (1):
- Research and Development Department, Medical School, Royal Derby Hospital, Derby, United Kingdom

REFERENCES:
- [Derived] Carter HM, Beard DJ, Leighton P, Moffatt F, Smith BE, Webster KE, Logan P. 'Going through the motions'; a rich account of the complexity of the anterior cruciate ligament reconstruction pathway, a UK qualitative study. BMJ Open. 2024 Sep 17;14(9):e079468. doi: 10.1136/bmjopen-2023-079468. PMID 39289010
- [Derived] Carter H, Beard D, Leighton P, Moffatt F, Smith BE, Webster KE, Logan P. Development of an intervention for patients following an anterior cruciate ligament rupture: an online nominal group technique consensus study. BMJ Open. 2024 Jul 18;14(7):e082387. doi: 10.1136/bmjopen-2023-082387. PMID 39025812

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - Preoperative: Interviews were completed with 18 participants who were at one of three time points on the patient pathway:
  1. Pre-anterior cruciate ligament surgery
  2. 3-month after anterior cruciate ligament surgery
  3. 12-months anterior cruciate ligament surgery
  Phase 1 - semi-structured interviews: Semi-structured face-to-face or virtual interviews.
- Phase 2 - Nominal Group Technique Panel: Consensus meetings were completed with 8 participants (clinicians, patients and stakeholders) to develop the intervention.
  Phase 2 - 2 online consensus meeting
Period: Overall Study
Arm/Group | Phase 1 - Preoperative | Phase 2 - Nominal Group Technique Panel
Started | 18 | 8
Completed | 18 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Preoperative | Phase 2 - Nominal Group Technique Panel | Total
Number analyzed (Participants) | 18 | 8 | 26
Age, Continuous [Median (Full Range); unit: years] | 29 [18 to 45] | NA [NA to NA] — Age note collected in phase 2 | NA [NA to NA] — Age note collected in phase 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | NA — Sex not collected for phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 15 | NA — Sex not collected for phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | NA — Ethnicity not collected in phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Indian | 2 | NA — Ethnicity not collected in phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
  British Asian | 1 | NA — Ethnicity not collected in phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Pakistani | 1 | NA — Ethnicity not collected in phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
Time-point on the pathway [Count of Participants; unit: Participants]
  Preoperative | 10 | NA — Not applicable to phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
  3-months post-operative | 6 | NA — Not applicable to phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
  12-months postoperative | 2 | NA — Not applicable to phase 2 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Semi-structured Interviews
Description: Understanding of patients' lived experiences of the treatment pathway following a diagnosis of an ACL rupture and agreed surgical management. Qualitative data collected from individual semi-structured interviews.
Time Frame: Interviews completed within approximately 60 minutes
Population: All participants remained in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Preoperative | Phase 2 - Nominal Group Technique Panel
Number analyzed (Participants) | 18 | 0
Participants
  Explore patient experiences of preoperative treatment | 18 | 0
  Explore patient experiences of postoperative treatment | 8 |
  Explore views and involvement in prehabilitation | 12 |
  Explore sources and consistency of healthcare advice | 18 |

2. Primary Outcome: Number of Participants in the Nominal Group Technique Panel
Description: Intervention developed with clinicians, patients and stakeholders for use with patients awaiting anterior cruciate ligament reconstruction in the National Health Service (NHS). Consensus was determined through voting set at an 70% threshold.
Time Frame: Two online meetings completed, up to 2 hours on 2 days approximately 1-month apart.
Population: All participant data analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Preoperative | Phase 2 - Nominal Group Technique Panel
Number analyzed (Participants) | 0 | 8
Participants
  Patient participants | 0 | 2
  Clinician participants | 0 | 5
  Therapy manager participant | 0 | 1

ADVERSE EVENTS:
Time Frame: The CI monitored risks for participants for the duration of the study (phase 1, 4 months). All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for Phase 2.
Description: Phase 1 - The CI will be responsible for assessing and managing risk, reporting this to the TMG and TSC as appropriate. This will be assessed and collected during the interviews with no further follow-up.
  There are no known risks to participation in phase 2 and averse events were not recorded over a period of time.
Arm/Group | Phase 1 - Preoperative | Phase 2 - Nominal Group Technique Panel
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/0
Other Adverse Events (participants affected / at risk) | 0/18 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT05529511/Prot_SAP_000.pdf